CLINICAL TRIAL: NCT07291193
Title: Impact of Sex Hormones on Human Skin Immunity in Health and Hidradenitis Suppurativa
Brief Title: Impact of Sex Hormones on Human Skin Immunity in Health and Hidradenitis Suppurativa (SIAP)
Acronym: SIAP
Status: Not yet recruiting | Type: Observational
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-072; 2025-A00923-46 (Other: ID-RCB number)
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Skin Immunity
Keywords: Pregnancy; Maternal Immunity; Skin; Hormones; Single Cell; Spatial-Omics
MeSH Terms: interventions — Blood Specimen Collection; Skin Microbiome; Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Healthy - Pregnant women: Adult woman, not affected by Hidradenitis Suppurativa, pregnant in her third trimester
  Interventions: Procedure: Blood sample, skin microbiota and biopsy
- Healthy - Non-pregnant women: Adult woman, not affected by Hidradenitis Suppurativa
  Interventions: Procedure: Blood sample, skin microbiota and biopsy
- Healthy - Men: Adult men, not affected by Hidradenitis Suppurativa
  Interventions: Procedure: Blood sample, skin microbiota and biopsy
- Hidradenitis suppurativa - Pregnant women: Adult woman, affected by Hidradenitis Suppurativa, pregnant in her third trimester
  Interventions: Procedure: Blood sample, skin microbiota and biopsy
- Hidradenitis suppurativa - Non-pregnant women: Adult woman, affected by Hidradenitis Suppurativa
  Interventions: Procedure: Blood sample, skin microbiota and biopsy
- Hidradenitis suppurativa - Men: Adult men, affected by Hidradenitis Suppurativa
  Interventions: Procedure: Blood sample, skin microbiota and biopsy

INTERVENTIONS:
Procedure: Blood sample, skin microbiota and biopsy — Blood sample (maximum 40mL) Skin microbiota (collection of cells from the skin surface using a swab (non-invasive) Skin biopsy, in hormone-dependent areas and/or in a non-hormone-dependent areas

SUMMARY:
Sex hormones are major regulators of skin immunity. Pregnancy represents a unique physiological state of profound hormonal remodeling. In late pregnancy, maternal levels of estrogens, progesterone, and other hormones increase dramatically, offering an unparalleled model to study the impact of sex hormones on skin immunity. Hidradenitis suppurativa (HS) provides a clinically relevant model to examine how sex hormones modulate skin inflammation.

DETAILED DESCRIPTION:
Sex hormones are major regulators of skin immunity. Recent work from Belkaid's laboratory in mice demonstrated that testosterone negatively regulated skin innate lymphoid cells (ILC2), leading to a reduction in dendritic cell accumulation and decreased activation in males, along with reduced tissue immunity. These findings highlight that sex-related differences in skin immunity emerge primarily after sexual maturation, driven by fluctuating hormone levels. However, whether these mechanisms are conserved in humans remains unknown.

Pregnancy represents a unique physiological state of profound hormonal remodeling. In late pregnancy, maternal levels of estrogens, progesterone, and other hormones increase dramatically, offering an unparalleled model to study the impact of sex hormones on skin immunity. Understanding maternal skin immunity is of particular importance, as the maternal immune system must balance tolerance to the fetus with protection against pathogens. Perturbation in this balance can have lasting effects on both maternal and child health. Faced with the dramatic increase in inflammatory and autoimmune disorders affecting children globally, understanding maternal immunity is of fundamental importance.

Hidradenitis suppurativa (HS) provides a clinically relevant disease model to examine how sex hormones modulate skin inflammation. HS is a chronic inflammatory skin disease with strong sex dimorphism: it affects predominantly women (70%) in Europe but is often more severe in men. In women, HS severity varies with the menstrual cycle and is frequently altered during pregnancy, suggesting a hormonal component in disease modulation. Yet, the mechanisms linking sex hormones, pregnancy, and skin immune responses in HS remain unexplored.

By systematically comparing men, non-pregnant women, and pregnant women, in both health and HS, this study will map immune cell populations in the skin and determine how sex hormones; testosterone, estrogens, and progesterone; shape cutaneous immunity at steady state and during inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Common criteria :
* Subject>18 years and <45 years,
* Written informed consent of the subject,
* Subject affiliated to the Assurance Maladie (French Health System) except Aide Médicale d'Etat (French State Medical Aid),
* Subject agrees that genomic analyses may be carried out on the samples
* Specific criteria :
* For pregnant women:Third trimester of pregnancy (between 29-37 weeks of amenorrhea).
* For HS subjects: Subject with hidradenitis suppurativa lesions at the sampling sites.

Exclusion Criteria:

* Common criteria :
* Subject immunocompromised,
* Subject under legal protection (guardianship or curatorship),
* Subject is unable to provide informed consent and to comply with the study requirements due to geographical, social, or psychiatric reasons,
* Subject in other research whose procedures may influence the immune system,
* Contraindication to any of medications listed in section 5.1 (antiseptic and local anesthetic used for biopsy(ies)),
* Subject whose health condition does not permit participation in study procedures.
* Specific criteria :
* For no HS subjects : Scarred skin at the biopsy site, Subject with pre-existing and/or still active inflammatory skin conditions, Subject experiencing early menopause (women) or andropause (men).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: As part of this study, adults (pregnant women, non-pregnant women, and men), healthy (not affected by HS) and affected by HS, will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of sex hormones and pregnancy on skin immunity by comparing immune cell populations in different populations (pregnant women, non-pregnant women, and men) with or without hidradenitis suppurativa. | 4 years
  Percentage of key skin immune cells (ILC2, dendritic cells, Langerhans cells), according to sex, pregnancy, and pathological context (healthy vs HS).

SECONDARY OUTCOMES:
Defining the spatial organisation of skin cells in order to assess how pregnancy remodels cutaneous immune responses in health and HS inflammation. | 4 years
  Immune cell mapping in healthy vs. inflamed skin biopsies across hormonal states (e.g. pregnancy).
Exploring how sex hormones, which are massively increased during pregnancy, and circulating immune profiling impact skin function and immunity. | 4 years
  Measurement of sex hormones and composition of PBMCs (Peripheral Blood Mononuclear Cells) in the blood of pregnant women and in controls (men and non-pregnant women).
Revealing the influence of the skin microbiota on the host immune system adapting to pregnancy in healthy and HS conditions. | 4 years
  Skin microbial metatranscriptomic profiling at the latest stage of pregnancy and in controls (men and non-pregnant women) in healthy and HS conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte OULES, MD-PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris